CLINICAL TRIAL: NCT00259480
Title: Reducing Family Caregiver Upset With Disruptive Behavior
Brief Title: Project ACT: Advancing Caregiving Techniques
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: R01AG022254 (NIH)
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Investigator

INTERVENTIONS:
Behavioral: Home Based Intervention — occupational therapy

SUMMARY:
The specific aims of this study are to:

1. Test the immediate effectiveness of the intervention to reduce caregiver upset with targeted disruptive behaviors (primary outcome). Hypothesis: Caregivers in the intervention group will report less upset with target behaviors at 4-months in comparison to caregivers in the control group.
2. Test the immediate effectiveness of the intervention to reduce caregiver burden (secondary outcome). Hypothesis: Caregivers in the intervention group will report less burden at 4-months in comparison to caregivers in the control group.
3. Test the immediate effectiveness of the intervention to reduce the frequency of occurrence of targeted disruptive behaviors in persons with dementia (secondary outcome). Hypothesis: Caregivers in the intervention group will report a decrease in the frequency of occurrence of targeted behaviors at 4-months in comparison to caregivers in the control group.
4. Test the maintenance effect of intervention at 6-months on caregiver upset and burden and targeted disruptive behaviors. Hypothesis: Compared to usual care, caregivers in intervention will maintain reduced upset and burden and report less occurrences of targeted behaviors from 4 to 6-months.
5. Assess the cost of the intervention and its cost effectiveness.

We have also received funding to conduct a supplementary study to evaluate the effect of the nurse intervention on behavior reduction and caregiver distress. The specific aims of this supplementary study arm are to: 1) describe the prevalence and type of medical conditions among control group participants who receive the nurse intervention, 2) describe for those with a detected medical condition/problem, the number of caregivers who follow-up with physicians and the type of physician follow-up/treatment that occurs; 3) evaluate whether control group participants who receive the nurse intervention report reduced disruptive behaviors and caregiver upset at 6 weeks (pre-post comparison); and 4) for control group participants who receive the nurse intervention, compare the level of disruptive behaviors and caregiver upset 4 months from entry into this study arm with the results in the Project ACT experimental group (who received the multi-component intervention).

ELIGIBILITY:
Inclusion Criteria:

* Caregivers are eligible for study participation if they:

  * are a family member 21 years of age or older (male or female),
  * live with the care recipient,
  * able to participate in the interview in English
  * have a telephone in their home,
  * plan to live in the area for 6 months, and
  * report a high level of upset with behaviors as follows. We will use the Agitated Behavior in Dementia Scale (ABID),62 which is a 16-item psychometrically valid scale of behavioral occurrences and associated caregiver upset. We chose this scale out of the six primary scales used to measure behavior given that the behaviors most closely match the intent of the intervention we plan to test. The behaviors include those listed earlier plus one additional behavior, repetitive vocalization. For each of these 17 behaviors that occur in the past week (for the purposes of screening eligibility, we will use a yes/no response format), caregivers are asked their level of upset (0 = not at all, 1 = a little, 2 = moderately, 3 = very much and 4 = extremely).
* Caregivers will be considered eligible if they obtain a total summed score of "3" or higher using the following algorithm:

  * Caregivers must report at least one behavior as very ("3") or extremely ("4") upset, or
  * caregivers must report three or more behaviors in which one behavior causes at least moderate ("2") level upset and one behavior causes at least a little upset.

Thus, caregivers with only scores of "1" ( a little upset) with three or more behavioral occurrences will not be considered eligible for this study. That is, this criteria excludes caregivers with no upset or a little upset. We will also require that the care recipient: 1) has a NINCDS-ADRDA diagnosis (physician generated) of dementia or a Mini-mental State Examination (MMSE) score of <23.

Exclusion Criteria:

* A caregiver is excluded if the caregiver or care recipient:

  * has a terminal illness with life expectancy < 6 months,
  * is in active treatment for cancer, or
  * has had >3 acute medical hospitalizations in the past year.
* Caregivers will also be excluded if:

  * they are currently involved in another clinical trial of psychosocial or educational interventions for caregivers; or
  * they are planning to place their family member in a nursing home within the next 6-months.
* Care-recipients will also be excluded if:

  * they have schizophrenia or a bi-polar disorder,
  * their dementia is secondary to probable head trauma,
  * their MMSE score = 0 and they are considered bed-bound, defined as confinement to bed or chair for at least 22 hours a day for at least four of the previous seven days,
  * a nursing home admission is planned to occur within six months or
  * they are enrolled in a clinical trial of pharmacological treatment for agitation.

These criteria exclude caregivers of ADRD patients at the severe stage of the disease process who may not benefit from the proposed intervention.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2001-08; Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Caregiver upset | Baseline, t2, t3
Care recipient behaviors | Baseline, t2, t3

SECONDARY OUTCOMES:
Caregiver self-efficacy | Baseline, t2, t3
Nursing home placement | When needed
Caregiver depression | Baseline, t2, t3

CONTACTS AND LOCATIONS:
Overall Officials: Laura N Gitlin, Ph.D, Principal Investigator — Thomas Jefferson University
Locations (1):
- Laura N. Gitlin,Ph.D, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Regier NG, Taylor JL, Szanton SL, Parmelee PA, Perrin N, Liu M, Jenkins E, Hodgson NA, Gitlin LN. Pain in persons with dementia and the direct and indirect impacts on caregiver burden. Geriatr Nurs. 2021 Mar-Apr;42(2):366-371. doi: 10.1016/j.gerinurse.2021.01.007. Epub 2021 Feb 8. PMID 33571930
- [Derived] Leggett AN, Kales HC, Gitlin LN. Finding fault: Criticism as a care management strategy and its impact on outcomes for dementia caregivers. Int J Geriatr Psychiatry. 2019 Apr;34(4):571-577. doi: 10.1002/gps.5052. Epub 2019 Jan 3. PMID 30556172
- [Derived] Rose KC, Gitlin LN. Background characteristics and treatment-related factors associated with treatment success or failure in a non-pharmacological intervention for dementia caregivers. Int Psychogeriatr. 2017 Jun;29(6):1005-1014. doi: 10.1017/S1041610217000205. Epub 2017 Mar 6. PMID 28260539
- [Derived] Gitlin LN, Rose K. Impact of caregiver readiness on outcomes of a nonpharmacological intervention to address behavioral symptoms in persons with dementia. Int J Geriatr Psychiatry. 2016 Sep;31(9):1056-63. doi: 10.1002/gps.4422. Epub 2016 Feb 2. PMID 26833933
- [Derived] Hodgson NA, Gitlin LN, Winter L, Czekanski K. Undiagnosed illness and neuropsychiatric behaviors in community residing older adults with dementia. Alzheimer Dis Assoc Disord. 2011 Apr-Jun;25(2):109-15. doi: 10.1097/WAD.0b013e3181f8520a. PMID 20921879